CLINICAL TRIAL: NCT04731974
Title: The Effectiveness of Melatonin for the Treatment of Acute Pediatric Concussion
Brief Title: Acute Concussion and Melatonin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Jeremy Root, Assistant Professor of Pediatrics and Emergency Medicine, George Washington Univ School of Medicine, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00015567
Record Dates: First submitted 2021-01-20; First posted 2021-02-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Concussion, Mild; Concussion, Brain; Pediatric ALL
MeSH Terms: conditions — Brain Concussion; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: This is a prospective single blinded randomized control trial of pediatric patients in the emergency department (ED) diagnosed with an acute concussion.
  Group A: melatonin Group B: routine/standard care
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Liquid Placebo
  Interventions: Other: Placebo
- Melatonin (Active Comparator): Liquid Melatonin
  Interventions: Drug: Melatonin 3 MG

INTERVENTIONS:
Drug: Melatonin 3 MG — Participants in the melatonin group will be instructed to take 3-mg liquid melatonin pill 1 hour prior to their habitual fall asleep time daily for 30 days.
  Arms: Melatonin
Other: Placebo — Participants in the placebo group will be instructed to take liquid placebo pill 1 hour prior to their habitual fall asleep time daily for 30 days.
  Arms: Placebo

SUMMARY:
In this study, the investigator plans a randomized trial of melatonin versus placebo post acute pediatric concussion. The investigator hypothesizes that patients with acute concussions managed with melatonin will have improved sleep, decreased depressive symptoms, decreased risk of prolonged concussion symptoms and faster resolution of concussion symptoms.

DETAILED DESCRIPTION:
To compare the risk of persistent post-concussive symptoms (PPCS) between melatonin and placebo after an acute pediatric concussion.

To determine if melatonin compared to placebo reduces the risk of PPCS for pediatric patients.

This is a prospective single-blinded randomized control trial of pediatric patients in the emergency department (ED) diagnosed with an acute concussion. Patients 12-18 years old with an acute concussion diagnosis will be eligible. All participants will receive actigraphy watches to wear on their wrists and measure sleep and activity patterns. Participants in the melatonin group will be instructed to take 3 mg of liquid melatonin 1 hour prior to their habitual fall asleep time daily for 30 days. Participants in the placebo group will be instructed to take their placebo liquid 1/2 hour prior to their habitual fall asleep time daily for 30 days.

All participants will be given standardized weekly assessments to track their concussion, sleep and depressive symptoms for one month. Research assistants will also arrange follow up in the telemedicine neurology headache clinic within 4 weeks post injury. At the follow-up visit, subjects will complete the Post Concussion Symptom Inventory (PCSI), Pediatric Sleep Disturbance (PSD), and Revised Childhood Anxiety and Depression Scales (RCADS).

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with an acute concussion within 72 hours
* Patient greater than 8 and less than 19 years old

Exclusion Criteria:

* Currently taking psychiatric medication
* Cognitive delay
* Glasgow Coma Score < 14
* positive findings on head computed tomography
* Any patient with intracranial surgery, pathology or instrumentation (e.g. ventriculoperitoneal shunt, brain tumor etc)
* Use of melatonin within the last week

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 254 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of average daily sleep duration between melatonin and placebo post acute pediatric concussion | 28 days post Emergency Department visit
  It is hypothesized that subjects managed with melatonin post an acute concussion will have increased sleep duration compared to placebo
Change in sleep quality between melatonin and placebo post acute pediatric concussion | 28 days post Emergency Department visit
  It is hypothesized that subjects managed with melatonin post an acute concussion will have increased sleep quality compared to placebo
Change in depressive symptoms between melatonin and placebo post acute pediatric concussion | 28 days post Emergency Department visit
  It is hypothesized that subjects managed with melatonin post an acute concussion will have decreased depressive symptoms compared to placebo

SECONDARY OUTCOMES:
Risk of persistent post-concussive symptoms between melatonin and placebo post acute pediatric concussion | 28 days post Emergency Department visit
  It is hypothesized that subjects managed with melatonin post an acute concussion will have a decreased relative risk of PPCS compared to those managed with placebo
Time to resolution of concussion symptoms between melatonin and placebo post acute pediatric concussion | 28 days post Emergency Department visit
  It is hypothesized that subjects managed with melatonin post an acute concussion will have a decreased time to resolution of concussion symptoms compared to those managed with placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
For the study, researchers will collect the age, sex, past medical history and through surveys, past, present and future symptoms after a head injury. This information will be used to determine which age groups are at risk and which constellation of symptoms persist following an acute head injury. All research documents and protected health information will be kept in a locked cabinet and a password protected RedCap database that only study staff personnel have access to. No data will be shared until manuscript is written, but will only be shared in manuscript and not in individual data. If significant adverse data is found for a patient, the Lead principal investigator will discuss with the subject and primary care physician.

REFERENCES:
- [Background] Barlow KM, Brooks BL, Esser MJ, Kirton A, Mikrogianakis A, Zemek RL, MacMaster FP, Nettel-Aguirre A, Yeates KO, Kirk V, Hutchison JS, Crawford S, Turley B, Cameron C, Hill MD, Samuel T, Buchhalter J, Richer L, Platt R, Boyd R, Dewey D. Efficacy of Melatonin in Children With Postconcussive Symptoms: A Randomized Clinical Trial. Pediatrics. 2020 Apr;145(4):e20192812. doi: 10.1542/peds.2019-2812. Epub 2020 Mar 26. PMID 32217739